CLINICAL TRIAL: NCT05849961
Title: TM-2023-017318 Exactech Hip Systems PMCF: A Post-Market Domestic (US) and International Data Collection to Assess Exactech Hip Systems
Brief Title: Exactech Hip Systems Post-Market Clinical Follow-up (PMCF)
Status: Recruiting | Type: Observational
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Other Study IDs: TM-2023-017318
Record Dates: First submitted 2023-04-14; First posted 2023-05-09 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Hip Arthroplasty, Total

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Prospective Subjects: Enrolled in the study pre-surgery. Subjects who agree to participate in the study that have not had surgery prior to being enrolled in the study.
  Interventions: Device: Exactech Hip Systems
- Retrospective to Prospective: Subjects enrolled in the study post- surgery then continue to participate in the study prospectively. Subjects who agree to participate in the study that have undergone surgery prior to enrollment in the study. Data for these subjects will collected from the subject's medical record for the time period prior to enrollment in the study containing data pertaining to the index surgery (retrospective data) and from the patient after they are enrolled in the study during the post-operative time period (prospectively).
  Interventions: Device: Exactech Hip Systems
- Retrospective Only Subjects: Subjects enrolled in the study post-study surgery with no intent to continue as prospective subjects. Patient's clinical record includes a signed HIPAA waiver allowing for the use of clinical record data for the purpose of clinical research outside of the operating institution.
  Interventions: Device: Exactech Hip Systems

INTERVENTIONS:
Device: Exactech Hip Systems — The Exactech Hip System comprises a fixed-bearing hip joint prostheses used in treating human hip joint diseases as part of THA. These prostheses include a combination of the components and are available in a range of sizes to accommodate varying anatomical requirements.

SUMMARY:
A Post-Market Domestic (US) and International Data Collection to Assess Exactech Hip Systems

DETAILED DESCRIPTION:
Patient outcomes data is important for assessing the post-market safety and effectiveness of orthopedic medical devices. The purpose of this study is to collect clinical and patient outcomes and survivorship data for patients who have received or will receive an Exactech Hip System for total hip arthroplasty (THA) prosthesis manufactured or distributed by Exactech Inc (Gainesville, Florida, USA).

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

* Subjects who agree to participate in the study that have not had surgery prior to being enrolled in the study.
* Skeletally mature (18 years of age or older).
* The subject is willing and able to provide written informed consent for participation in the study.
* Subject is to receive an Exactech Hip System THA for any approved indication for use.
* The hip replacement will be performed by the investigator or a surgeon sub- investigator.
* The devices will be used according to the approved indications.

Cohort 2:

* Subjects who agree to participate in the study that have undergone surgery prior to enrollment in the study. Data for these subjects will be collected from the subject's medical record for the time-period prior to enrollment in the study containing data pertaining to the preoperative time period and index surgery (retrospective data) and from the patient after they are enrolled in the study during the post-operative time- period (prospectively).
* Skeletally mature (18 years of age or older).
* The subject is willing and able to provide written informed consent for participation in the study.
* Subject received an Exactech Hip System THA for any approved indication for use.
* The hip replacement was performed by the investigator or a surgeon sub-investigator.
* The devices are/were used according to the approved indications.
* Special consideration should be taken to ensure that these subjects meet all inclusion criteria, none of the exclusion criteria, and have a minimum of the following pre- operative, operative, and applicable postoperative data available in the subject's medical records, related to the Exactech Hip System prosthesis manufactured or distributed by Exactech Inc (Gainesville, Florida, USA). Prior to inclusion in the study, the following details must be available for data submission:

Pre-Operative:

Demographic Data

* Gender
* Age at surgery
* Height/Weight
* Indication for surgery
* Prior Injuries/Surgeries on index hip
* Comorbidities

Operative:

* Date of Surgery
* Type of Surgery (Primary / Revision)
* All component product information, including catalogue reference numbers.
* Adverse Event Information, if applicable

Cohort 3:

Note: No prospective data may be collected from a subject if they are enrolled under this cohort unless the subject is willing and able to provide written informed consent for participation in the study, in which case they should be part of Cohort 2.

* Skeletally mature (18 years of age or older).
* The subject is willing and able to provide written informed consent for participation in the study.
* Subject received an Exactech Hip System THA for any approved indication for use.
* The hip replacement was performed by the investigator or a surgeon sub-investigator.
* The devices are/were used according to the approved indications.
* Special consideration should be taken to ensure that these subjects meet all inclusion criteria, none of the exclusion criteria, and have a minimum of the following pre- operative, operative, and applicable postoperative data available in the subject's medical records, related to the Exactech Hip System prosthesis manufactured or distributed by Exactech Inc (Gainesville, Florida, USA). Prior to inclusion in the study, the following details must be available for data submission:

Pre-Operative:

Demographic Data

* Gender
* Age at surgery
* Height/Weight
* Indication for surgery
* Prior Injuries/Surgeries on index hip
* Comorbidities

Operative:

* Date of Surgery
* Type of Surgery (Primary / Revision)
* All component product information, including catalogue reference numbers.
* Adverse Event Information, if applicable

Exclusion Criteria:

* Patient was <18 years of age at time of surgery
* Patient does not meet the indicated population for use criteria for this device.
* Patient is pregnant
* Patient is a prisoner
* Patient has a physical or mental condition that would invalidate the results
* Patient is contraindicated for the surgery (e.g., metal allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must qualify for surgery per indications and contraindications and meet all the inclusion criteria and none of the exclusion criteria. The decision to offer a patient enrollment in this study is left to the surgeon's discretion.
Sampling Method: Non-Probability Sample
Enrollment: 2946 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2036-07-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score | Preoperative
  Harris Hip Score (HHS) - validated outcome score. Scores range from 0 (worse disability) to 100 (less disability). The HHS will be collected throughout the duration of the implanted device according to standard of care.
Harris Hip Score | 4-6 week Post-op; per standard of care
  Harris Hip Score (HHS) - validated outcome score. Scores range from 0 (worse disability) to 100 (less disability). The HHS will be collected throughout the duration of the implanted device according to standard of care.
Harris Hip Score | 3-6 month Post-op; per standard of care
  Harris Hip Score (HHS) - validated outcome score. Scores range from 0 (worse disability) to 100 (less disability). The HHS will be collected throughout the duration of the implanted device according to standard of care.
Harris Hip Score | Annually up to 10 years; per standard of care
  Harris Hip Score (HHS) - validated outcome score. Scores range from 0 (worse disability) to 100 (less disability). The HHS will be collected throughout the duration of the implanted device according to standard of care.
Oxford Hip Score | Preoperative
  Oxford Hip Score (OHS) - validate outcome score. Scores range from score 0 (most severe symptoms, to 48 (least symptoms). The OHS will be collected throughout the duration of the implanted device according to standard of care.
Oxford Hip Score | 4-6 week Post-op; per standard of care
  Oxford Hip Score (OHS) - validate outcome score. Scores range from score 0 (most severe symptoms, to 48 (least symptoms). The OHS will be collected throughout the duration of the implanted device according to standard of care.
Oxford Hip Score | 3-6 month Post-op; per standard of care
  Oxford Hip Score (OHS) - validate outcome score. Scores range from score 0 (most severe symptoms, to 48 (least symptoms). The OHS will be collected throughout the duration of the implanted device according to standard of care.
Oxford Hip Score | Annually up to 10 years; per standard of care
  Oxford Hip Score (OHS) - validate outcome score. Scores range from score 0 (most severe symptoms, to 48 (least symptoms). The OHS will be collected throughout the duration of the implanted device according to standard of care.

CONTACTS AND LOCATIONS:
Locations (1):
- Tulsa Bone & Joint Associates, Tulsa, Oklahoma, United States